CLINICAL TRIAL: NCT06087250
Title: Reliability of Carotid Artery Corrected Flow Time Predicting Fluid Responsiveness in Geriatric Patients.
Brief Title: Carotid Artery Corrected Flow Time and Fluid Responsiveness in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Beliz Bilgili, Associated Prof, M.D, Marmara University
Other Study IDs: 2023
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Fluid Responsiveness; Common Carotid Artery
Keywords: fluid responsiveness; carotid blood flow; carotid corrected flow time

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fluid responsive: A 15% increase in cardiac output following a fluid challenge ( 6ml/kg crystalloid solution infusion in 30 min).
  Carotid corrected flow time measured before and after fluid challenge by ultrasound.
- Fluid non-responsive: Failure of 15% increase in cardiac output following a fluid challenge ( 6ml/kg crystalloid solution infusion in 30 min).
  Carotid corrected flow time measured before and after fluid challenge by ultrasound.

SUMMARY:
Carotid blood flow and corrected carotid flow time (Carotid Flow Time (FTc)) provide information about left ventricular preload and inversely correlate with systemic vascular resistance. The reliability in assessing fluid responsiveness has been demonstrated in studies involving invasive cardiac output measurements. In the elderly patient population where arterial elasticity can be compromised, there is no existing data in literature that determines the reliability and predictive value of FTc after general anesthesia induction.

DETAILED DESCRIPTION:
Doppler ultrasound of the common carotid artery has begun to be used as a potential non-invasive tool for assessing hemodynamic status. Its non-invasive nature, ability to be applied independently of the patient's position, ease of application due to the superficial location of the carotid artery, and resistance to intrathoracic pressure changes are among its advantages. Carotid blood flow and corrected carotid flow time (Carotid Flow Time (FTc)) provide information about left ventricular preload and inversely correlate with systemic vascular resistance. Additionally, the velocity time integral (VTI) measuring blood flow through the carotid artery during systole, when multiplied by the cross-sectional area of the carotid artery, allows for the determination of flow within the carotid artery. The reliability in assessing fluid responsiveness has been demonstrated in studies involving invasive cardiac output measurements. In the elderly patient population where arterial elasticity can be compromised, there is no existing data in literature that determines the reliability and predictive value of FTc after general anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* geriatric patient (older than 65 years of age) having surgery under general anesthesia

Exclusion Criteria:

* Common carotid artery stenosis, common carotid artery disease

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — older than 65 years of age
Study Population: geriatric patient (older than 65 years of age) having surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
carotid corrected flow time (cFT) | 1 hour
  the ability ofc FT to predict fluid responsiveness

SECONDARY OUTCOMES:
cutt-of value of cFT | 1 hour
  the cutt-of value of cFT to predict fluid responsiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)